CLINICAL TRIAL: NCT01302015
Title: Safety and Efficacy of Autologous Adipose Tissue Derived Mesenchymal Stem Cells Transplantation in Patient With Buerger's Disease
Brief Title: Autologous Adipose Tissue Derived Mesenchymal Stem Cells Transplantation in Patient With Buerger's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: R-Bio (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Vascostem
Record Dates: First submitted 2011-02-17; First posted 2011-02-23 (Estimated); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Buerger's Disease
MeSH Terms: conditions — Thromboangiitis Obliterans

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RNL-Vascostem® (Experimental): drug name and ingredients : RNL-Vascostem[Autologous adipose tissue derived mesenchymal stem cells] dosage : Intramuscular infusion, 5 x 10e6 cells/kg
  Interventions: Biological: RNL-Vascostem®

INTERVENTIONS:
Biological: RNL-Vascostem®
  Other Names: Autologous adipose tissue derived mesenchymal stem cells

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of autologous transplantation of Adipose Tissue derived Mesenchymal stem cells (MSCs) in patient with Buerger's disease.

DETAILED DESCRIPTION:
Buerger's disease, also known as thromboangiitis obliterans, is a rare disorder that, in most cases, affects young or middle-aged male cigarette smokers. It is characterized by narrowing or blockage (occlusion) of the veins and arteries of the extremities, resulting in reduced blood flow to these areas (peripheral vascular disease). The exact cause of Buerger's disease is not known; however, most affected individuals are heavy tobacco users.

This drug is an autologous cell treatment for necrosis in the legs of patients with Beurger's diseases to improve symptoms through vascular regeneration.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who understand and sign the consent form for this study.
* Age :20-80, males and females
* Patients at least 6 months after Buerger's disease
* Patients with a luminal stenosis of more than 50% on angiography
* Rutherford class II-4, III-5 or III-6
* Subjects not eligible to undergo a revascularization or vascular bypass graft
* Patients who can't treat with traditional medication and need a arthroplasty.
* Patients whose lesion is 2~6 cm2 in size
* Duration of pain over Grade 4(11-point numeric scale) : > 4 months

Exclusion Criteria:

* Subjects who cannot survive more than 6 months with critical other complications.
* Patient with well-known active malignant tumor.
* Patients who exceed normal reference values from following test : PAP smear screening, chest X-ray, PSA, mammogram, occult blood test
* Patients in need of a immediate amputation and have a potentially life-threatening complications of critical ischemia
* Patients with uncontrolled iliac artery obstruction of targeted areas.
* Condition with targeted lower limb that have widespread necrosis or in need of amputation.
* End-stage renal failure patients who depend on hemodialysis
* Patients with uncontrolled diabetes mellitus (HbA1c > 10%).
* Treatment with immunosuppressant (prednisone > 5mg/day).
* Treatment with a anti-inflammatory drugs within 1 weeks prior to enrollment.
* Women who are pregnant or breast feeding or planning to become pregnant during the study.
* Subjects who have cerebrovascular accident within 6 months prior to inclusion in the study.
* Patients with acute myocardial infarction, angina pectoris.
* Subjects who had been underwent a cardiovascular surgery such as carotid endarterectomy, arterial aneurysm, bypass surgery and coronary bypass surgery within 3 months prior to inclusion in the study.
* Participation in another clinical trial or treatment with a different investigational product within 3 months prior to inclusion in the study.
* Other pathologic conditions or circumstances that difficult participation in the study according to medical criteria

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2007-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Treadmill Walking Distance | 24 weeks
  Improvement in TWD(Treadmill Walking Distance)

SECONDARY OUTCOMES:
VAS(Visual Analog Scale) | 24 weeks
  Improvement in VAS(Visual Analog Scale) score
Toe-Brachial Pressure Index, TBPI | 24 weeks
  Improvement in TBPI score
Transcutaneous oxygen pressure, TcPO2 | 24 weeks
  Improvement in TcPO2 score
Arterial Brachial Pressure Index, ABPI | 24 weeks
  Improvement in ABPI score
Pain Free Walking Distance, PFWD | 24 weeks
  Improvement in PFWD score
Angiography | 24 weeks
  Improvement on Angiography
Laser Doppler | 24 weeks
  Improvement on Laser Doppler
dose and frequency in use of a analgesic medicine | 24 weeks
  Changes in dose and frequency in use of a analgesic medicine
Safety Evaluation | 24 weeks
  To determine the overall safety of RNL-VascoStem® carrier using physical examinations, vital signs, treatment emergent adverse events (TEAEs), and the results of clinical lab tests

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Hong Baek, M.D.&Ph.D., Principal Investigator — Seoul St. Mary's Hospital; Eui Cheol Jeong, M.D., Principal Investigator — SMG-SNU Boramae Medical Center
Locations (2):
- South Korea (2):
  - Seoul St. Mary's Hospital, Seoul
  - SMG-SNU Boramae Medical Center, Seoul

REFERENCES:
- [Result] Lee HC, An SG, Lee HW, Park JS, Cha KS, Hong TJ, Park JH, Lee SY, Kim SP, Kim YD, Chung SW, Bae YC, Shin YB, Kim JI, Jung JS. Safety and effect of adipose tissue-derived stem cell implantation in patients with critical limb ischemia: a pilot study. Circ J. 2012;76(7):1750-60. doi: 10.1253/circj.cj-11-1135. Epub 2012 Apr 12. PMID 22498564